CLINICAL TRIAL: NCT05410210
Title: A Randomized Controlled Trial to Study the Impact of Pharmaceutical Care on Drug-related Problems in Patients With Parkinson's Disease at Parkinson's Disease and Movement Disorders Clinic, Siriraj Hospital, Thailand
Brief Title: Impact of Pharmaceutical Care on Drug-related Problems in Patients With Parkinson's Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mahidol University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 1040/2564(IRB4) MOU
Record Dates: First submitted 2022-05-13; First posted 2022-06-08 (Actual); Last update posted 2023-10-10 (Actual); Status verified 2023-10

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease | interventions — Pharmaceutical Services

STUDY DESIGN:
Who Masked: Participant
Masking Description: The participants and assessors evaluating MDS-UPDRS were blinded in this study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pharmaceutical care (Experimental): The intervention group will receive the pharmaceutical care from a pharmacist and the existing standard care available in the Parkinson's disease and movement disorders clinic.
  Interventions: Other: Pharmaceutical care
- Usual care (No Intervention): The usual care includes the current existing care provided to patients in the Parkinson's disease and movement disorders clinic except the pharmaceutical care provided by pharmacists.

INTERVENTIONS:
Other: Pharmaceutical care — The clinical pharmacists will conduct medication reviews, patient education, and counseling. Moreover, the clinical pharmacists will identify drug-related problems (DRPs) and provide the information through written pharmacist notes to physicians at the clinic.
  Arms: Pharmaceutical care

SUMMARY:
The aim of this study is to evaluate the impact of pharmaceutical care on the number of drug-related problems, clinical outcomes and quality of life of patients with Parkinson's disease.

DETAILED DESCRIPTION:
This is a randomized controlled study that will be conducted in Parkinson's disease and movement disorders clinic, Siriraj Hospital, Thailand. The participants and assessors evaluating MDS-UPDRS were blinded in this study.

The participants will be divided into two groups by block randomization: intervention group and usual care group.

For the intervention group, the clinical pharmacists will conduct medication reviews, patient education, and counseling. Moreover, the clinical pharmacists will identify drug-related problems (DRPs) and provide the information through written pharmacist notes to physicians at the clinic. For patients randomized to the control group will attend the medical follow-up as usual and receive usual care. Telepharmacy will be conducted 2-7 days before the doctor visit and within 1 week after the doctor visit. Data collection will be conducted at baseline, week 12, and week 24 in both groups. After the follow-up, the pharmacist will count the number of drug-related problems identified after the doctor visit. The primary outcome of the study is comparing the number of drug-related problems per person changed from the start of the study to the end of week 24 between two groups.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years or older
2. Diagnosed with idiopathic Parkinson's disease according to the UK Parkinson's disease Society Brain Bank Criteria for at least 3 years
3. Modified Hoehn and Yahr stage 2-4
4. Patient had received at least one of antiparkinsonian drugs the following: levodopa, MAO-B inhibitors, dopamine agonists, COMT inhibitors, amantadine, and trihexyphenidyl
5. Patient has given a written informed consent to participate in the study. If the patients are unable to give an informed consent, it must be obtained from the caregiver.

Exclusion Criteria:

1. Patient is unable to communicate via telephone or mobile phone or internet.
2. Patient who is terminal illness
3. Patient who is bed ridden
4. Patient with other movement disorders include corticobasal syndrome, multiple system atrophy, progressive supranuclear palsy and essential tremor
5. Moderate to severe dementia as evidenced by Mini Mental State Examination (MMSE) or Thai Mental State Examination (TMSE) less than 20 and without the caregiver
6. Patient who is planning to undergo surgery or have a history of surgical treatment for Parkinson's disease such as pallidotomy, thalamotomy, or deep brain stimulation
7. Patient with hearing impairments which affects communication via telephone or electronic media
8. Unable to communicate Thai language

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2022-03-11 (Actual); Primary Completion 2022-12-02 (Actual); Study Completion 2023-01-23 (Actual)

PRIMARY OUTCOMES:
Change in the total number of drug-related problems related to all drugs | 24 weeks
  Compare the change of mean number of drug-related problems related to all drugs per person between the pharmaceutical care versus the usual care group.

SECONDARY OUTCOMES:
Change in the number of drug-related problems related to with Parkinson's disease treatment | 24 weeks
  Compare the change of mean number of drug-related problems with Parkinson's disease treatment per person between the pharmaceutical care versus the usual care group.
Change in clinical outcome | 12 and 24 weeks
  Clinical outcome is assessed using Movement Disorder Society-Unified Parkinson's Disease Rating Scale (MDS-UPDRS) scores. Compare the change in MDS-UPDRS scores (both total score and separate part) between the pharmaceutical care group and the usual care group. The minimum and maximum value are 0 and 199, respectively. The higher scores mean a worse outcome.
Clinical status | 12 and 24 weeks
  Clinical status is assessed using Patient Global Impression of Change (PGIC). Compare the mean scores of PGIC at 12 and 24 weeks between the pharmaceutical care group and the usual care group. The minimum and maximum value are 1 and 7, respectively. The higher scores mean a worse outcome.
Change in Quality of life | 24 weeks
  Quality of life is assessed using the 8-item version of the Parkinson's Disease Questionnaire (PDQ-8). Compare the change in PDQ-8 scores between the pharmaceutical care group and the usual care group. The minimum and maximum value are 0 and 32, respectively. The higher scores mean a worse outcome.
The factors affecting the change in the number of drug-related problems | 24 weeks
  ● The regression coefficient of the factors affecting the change in the number of drug-related problems were pharmaceutical care (yes/no), the number of drug-related problems at the start of the study (in items), the number of drug types the patient received at the start of the study (in items), disease duration (in years), and the Hoehn & Yahr stage (2-4)
The factors affecting the change in the PGIC | 24 weeks
  ● The regression coefficient of the factors affecting the change in the PGIC were pharmaceutical care (yes/no), the number of drug-related problems at the start of the study (in items), the number of drug types the patient received at the start of the study (in items), disease duration (in years), and the Hoehn & Yahr stage (2-4)

CONTACTS AND LOCATIONS:
Overall Officials: Yuvadee Pitakpatapee, Principal Investigator — Yuvadee.pit@gmail.com
Locations (1):
- Siriraj hospital, Bangkok, Thailand

REFERENCES:
- [Derived] Techa-Angkoon P, Pitakpatapee Y, Saengphatrachai W, Srivanitchapoom P, Suansanae T. Impact of pharmacist-physician collaboration on patient outcomes in Parkinson's disease: a randomised controlled trial in tertiary care. Int J Clin Pharm. 2025 Jun;47(3):834-843. doi: 10.1007/s11096-025-01883-6. Epub 2025 Feb 13. PMID 39945968